CLINICAL TRIAL: NCT00380367
Title: Evaluation of Safety, Tolerability and Immunogenicity of Quadrivalent HPV Vaccine in Healthy Females 9 to 15 Years of Age in India
Brief Title: Safety, Tolerability and Immunogenicity of HPV (Human Papilloma Virus) Vaccine in Healthy Females 9 to 15 Years of Age in India (V501-029)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V501-029; 2006_038 (Other: Merck Registration Number); 2017-000111-16 (EudraCT Number)
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Results first posted 2009-04-14 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quadrivalent HPV VLP Vaccine (Types 6, 11, 16, 18) (Experimental): Participants who enroll receive a total of 3 intramuscular injections of Quadrivalent HPV VLP vaccine (types 6, 11, 16, 18) given on Day 1, Month 2 and Month 6.
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine — Quadrivalent HPV vaccine (6, 11, 16, 18) given intramuscularly on Day 1, Month 2, and Month 6.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of the Quadrivalent Human Papilloma Virus (HPV) vaccine in healthy females 9 to 15 years of age in India. Quadrivalent HPV Vaccine is composed of L1 virus-like particles (VLPs) from HPV types 6, 11, 16, and 18.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Females Age 9 To 15 Years
* Females Not Sexually Active And Not Plan On Becoming Sexually Active During The Study
* No Fevers 24 Hours Prior To The First Injection

Exclusion Criteria:

* Participant Had Received A Prior Vaccination With A HPV Vaccine
* Participant Has Allergies To Vaccine Component Including Aluminum And Yeast
* Participant Has (Human Immunodeficiency Virus) HIV Infection
* Participant Is Immunocompromised
* Participant Received Or Plans To Receive Blood-Derived Product Within 6 Months Prior To The First Injection
* Participant Received Or Plans To Receive Immune Globulin Preparation Within 6 Months To The First Injection

Ages: 9 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2007-05-03 (Actual); Primary Completion 2008-02-04 (Actual); Study Completion 2008-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Garland SM, Anagani M, Bhatla N, Chatterjee S, Lalwani S, Ross C, Group T, Lin J, Luxembourg A, Walia A, Tu Y. Immunogenicity and safety of quadrivalent and 9-valent human papillomavirus vaccines in Indian clinical trial participants. Hum Vaccin Immunother. 2022 Nov 30;18(6):2105067. doi: 10.1080/21645515.2022.2105067. Epub 2022 Aug 23. PMID 35997582

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In (FPI): 03 May 2007 Last Patient Out (LPO): 04 Feb 2008
  Multi-center study. Seven sites participated in the study. All sites were medical centers located in Bangalore, Mumbai and Pune.
Pre-assignment Details: Open-label, single-arm, nonrandomized study. Females >9 to 15 years of age, who have not had coitarche and did not plan on becoming sexually active through the course of the study, who did not have a feverish feeling within 24 hours prior to the first injection, were included in the study.
Groups:
- Quadrivalent HPV VLP Vaccine (Types 6, 11, 16, 18): Participants who were enrolled received a total of 3 intramuscular injections of Quadrivalent Human Papilloma Virus (HPV) virus like particles (VLP) vaccine (types 6, 11, 16, 18) given on Day 1, Month 2 and Month 6.
Period: Overall Study
Arm/Group | Quadrivalent HPV VLP Vaccine (Types 6, 11, 16, 18)
Started | 110
Completed | 108
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Quadrivalent HPV VLP Vaccine (Types 6, 11, 16, 18)
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.54 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 16.76 (2.79)
Height [Mean (Standard Deviation); unit: Cm] | 143.32 (9.58)
Weight [Median (Standard Deviation); unit: Kg] | 34.90 (8.81)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Seroconvert to Each HPV Serotype (Types 6, 11, 16, 18) at Month 7
Description: Month 7 HPV competitive Luminex Immunoassay (cLIA) seroconversion rates among participants who received Quadrivalent HPV (Types 6, 11, 16, 18) Late 1 (L1) capsid protein VLP vaccine were reported. The quadrivalent HPV competitive cLIA (v2.0) was used to detect antibody to HPV VLPs serotypes 6, 11, 16, 18 before and after vaccination with the HPV quadrivalent vaccine. Seropositivity cutoffs of the HPV cLIAs were assessed using a panel of sera from participants highly likely to be HPV naïve (children), and from participants who were highly likely to be seropositive. Any sample with a value less than the cutoffs was considered serostatus negative. Samples with values equal to or greater than the cutoff were considered serostatus positive. The cutoffs for the HPV 6, 11, 16, and 18 cLIAs were 20 milli-Merck units per milli liter (mMU/mL), 16 mMU/mL, 20 mMU/mL, and 24 mMU/mL, respectively.
Time Frame: One month post-dose 3 (Month 7)
Population: Per-Protocol (P-P) immunogenicity population: All participants who were not general protocol violators, received all 3 vaccinations within acceptable day ranges, were sero-negative at Day 1 for the relevant HPV type(s), and had a Month 7 serum sample collected within an acceptable day range.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Quadrivalent HPV VLP Vaccine (Types 6, 11, 16, 18)
Number analyzed (Participants) | 105
percentage of participants
  Anti-HPV 6 (n=99) | 96.97 [93.59 to 100.35]
  Anti-HPV 11 (n=105) | 99.05 [97.19 to 100.91]
  Anti-HPV 16 (n=105) | 99.05 [97.19 to 100.91]
  Anti-HPV 18 (n=105) | 99.05 [97.19 to 100.91]

2. Primary Outcome: Number of Participants With Any Adverse Events (AEs), Injection-site AEs, Systemic AEs, or Vaccine-related AEs During the Study
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the SPONSOR's product, was also an AE. Pre-specified injection site AEs included pain, tenderness, erythema, and swelling. A vaccine-related AE was an AE considered by the investigator to be possibly, probably, or definitely related to the vaccine. All AEs collected on participant's Vaccination Report Card daily for 14 days after each vaccination (Days 1-15).
  The number of participants who experienced ≥1 AE, the number of participants who experienced ≥1 injection site AE, the number of participants who experienced ≥1 systemic AE, and the number of participants who experienced ≥1 vaccine-related AE were reported for the Safety Cohort.
Time Frame: Up to 7 months
Population: Safety Cohort: All enrolled participants who received ≥1 injection and had safety follow-up data. Two participants did not have safety follow-up data and were excluded from safety analyses.
Measure: Number; unit: participants
Arm/Group | Quadrivalent HPV VLP Vaccine (Types 6, 11, 16, 18)
Number analyzed (Participants) | 108
participants
  Any AE | 63
  Injection site AE | 50
  Systemic AE | 35
  Vaccine-related AE | 45

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: Safety Cohort: All enrolled participants who received ≥1 injection and had safety follow-up data. Two participants did not have safety follow-up data and were excluded from safety analyses.
Arm/Group | Quadrivalent HPV VLP Vaccine (Types 6, 11, 16, 18)
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 63/108
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent HPV VLP Vaccine (Types 6, 11, 16, 18) (N=108)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Flank pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 25 (25)
Nasopharyngitis (Infections and infestations) | 8 (8)
Pharyngitis (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Somnolence (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Injection site pain (General disorders) | 46 (83)
Injection site tenderness (General disorders) | 25 (41)
Injection site erythema (General disorders) | 13 (20)
Injection site swelling (General disorders) | 10 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.